CLINICAL TRIAL: NCT00884689
Title: A 6 Months NIS to Evaluate the Use of Rescue Medication and Quality of Life in Adult Asthmatic Subjects Treated With Symbicort® SMART® 1-2 Inhalations b.i.d. as Maintenance Therapy Plus Additional Inhalations As-needed, Compared to Patients Treated With a Free Combination of an Inhaled Glucocorticosteroid and an Inhaled Long Acting ß2-agonist Plus as Needed Inhalations of a Short Acting ß2 Agonist.
Brief Title: A 6 Months NIS to Evaluate the Use of Rescue Medication and Quality of Life in Adult Asthmatic Subjects Treated With Symbicort® SMART®
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: ClinResearch, GmbH (Other)
Responsible Party: Dr. Kai Richter, Vice President Medical
Other Study IDs: NIS-RDE-SYM-2009/1
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Asthma
Keywords: Symbicort SMART; Free Combination GCS/LABA treatment
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Asthma patient with specific treatment
- 2: Asthma patient on different specific treatment compared to the other group

SUMMARY:
The purpose of this study is to describe the use of rescue medication and quality of life in adult asthmatic patients, either treated with SYMBICORT SMART® (regular dose according to physician's prescription and the current summary of product characteristics - SPC) or treated with a free combination of ICS plus LABA plus as needed SABA prescribed by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of asthma demonstrating a reversible obstruction during the last 5 years prior to visit 1.
* Patients being prescribed either Symbicort SMART or a free combination of ICS and LABA with SABA as rescue inhaler and being on that treatment for at least 3 month.
* A history (documented in the patient's file) of at least one severe asthma exacerbation within 24 months prior to visit 1 but not within the last 30 days prior to Visit 1.
* A severe asthma exacerbation is defined as a deterioration of asthma leading to at least one of the following:

  * Oral/systemic GCS treatment due to asthma for at least 3 days
  * Unscheduled health-care visit due to asthmaHospitalization or emergency room visit because of asthma requiring treatment with oral/systemic GCS

Exclusion Criteria:

* Intake of oral, rectal, or parenteral GCS within 30 days prior to visit
* Use of ß-blocking agents
* Respiratory infection affecting the asthma, as judged by the investigator, within 30 days prior to visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma treatment will not be assigned randomly, but will be administered at the discretion of the physicians according to standard medical practice. Each site should enrol 5 patients using the Symbicort® SMART® principle and 5 patients being prescribed a free combination GCS / LABA treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-04; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Use of rescue medication | daily during 6 month

SECONDARY OUTCOMES:
Quality of life | 3 times during study
Efficacy variables | during 6 month
Safety variables | during 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Kai Richter, MD, Study Director — AstraZeneca
Locations (43):
- Germany (43):
  - Research Site, Aschaffenburg
  - Research Site, Bad Lippspringe
  - Research Site, Bad Sassendorf
  - Research Site, Bergkamen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Braunschweig
  - Research Site, Buchholz
  - Research Site, Chemnitz
  - Research Site, Coswig
  - Research Site, Cottbus
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Frankfurt
  - Research Site, Fürth
  - Research Site, Gelsenkirchen
  - Research Site, Gütersloh
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Ketzin
  - Research Site, Köthen
  - Research Site, Leipzig
  - Research Site, Löhne
  - Research Site, Lübeck
  - Research Site, Lüdenscheid
  - Research Site, Marburg
  - Research Site, Marl
  - Research Site, Mittelbach
  - Research Site, Mühlhausen
  - Research Site, Mülheim
  - Research Site, München
  - Research Site, Oschersleben
  - Research Site, Potsdam
  - Research Site, Remscheid
  - Research Site, Saarlouis
  - Research Site, Schwetzingen
  - Research Site, Steinhagen
  - Research Site, Stockach
  - Research Site, Wedel
  - Research Site, Wesseling
  - Research Site, Weyhe